CLINICAL TRIAL: NCT02291848
Title: Administration of Tumor-Associated Antigen (TAA)-Specific Cytotoxic T-Lymphocytes to Patients with Active Myeloma (TACTAM)
Brief Title: Tumor-Associated Antigen-Specific Cytotoxic T-Lymphocytes for Multiple Myeloma
Acronym: TACTAM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); Harris County Hospital District (Other Government)
Responsible Party: Principal Investigator, Premal Lulla, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35626, TACTAM
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cytotoxic T-lymphocytes
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Patients receiving TAA-specific CTLs as therapy for Myeloma
  Interventions: Biological: TAA-specific CTLs
- Group B (Experimental): Patients receiving TAA-Specific CTLs as adjunctive therapy following autologous or syngeneic transplant for myeloma
  Interventions: Biological: TAA-specific CTLs
- Group C (Experimental): Patients with high risk MGUS or smoldering myeloma receiving a fixed dose TAA-Specific CTLs
  Interventions: Biological: TAA-specific CTLs- fixed dose

INTERVENTIONS:
Biological: TAA-specific CTLs — Groups A and B only: Each patient will receive 2 infusions at the same dose, 14 days apart, according to the following dosing schedules:
  Dose Level One:
  Day 0: 5 x 10^6 cells/m2 and Day 14: 5 x 10^6 cells/m2
  Dose Level Two:
  Day 0: 1 x 10^7 cells/m2 and Day 14: 1 x 10^7 cells/m2
  Dose Level Three:
  Day 0 2 x 10^7 cells/m2 and Day 14 2 x 10^7 cells/m2
  If patients without measurable disease remain in complete remission or those patients with measurable active disease (for multiple myeloma, MGUS or smoldering myeloma) at the time of infusion have stable disease or a partial response at their 8 week or subsequent evaluations, they are eligible to receive up to 6 additional doses of CTLs at monthly intervals-each of which will consist of the same cell number or less (if there is not enough product) than their second infusion.
  Arms: Group A; Group B
Biological: TAA-specific CTLs- fixed dose — Fixed dose of 2 infusions of 2 x 10^7 cells/m2 administered 2 weeks apart.
  If patients without measurable disease remain in complete remission or those patients with measurable active disease (for multiple myeloma, MGUS or smoldering myeloma) at the time of infusion have stable disease or a partial response at their 8 week or subsequent evaluations, they are eligible to receive up to 6 additional doses of CTLs at monthly intervals-each of which will consist of the same cell number or less (if there is not enough product) than their second infusion.
  Arms: Group C

SUMMARY:
This study is for patients that have a cancer called Multiple Myeloma, monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SM). MGUS and SM have tumor cells that possess nearly identical properties to the cancer cells seen in patients with multiple myeloma.

The investigators would like to target proteins that are expressed by these cells using the patient's own immune cells known as T lymphocytes.This research study uses special immune system cells called tumor associated antigen (TAA)-specific cytotoxic T lymphocytes (CTLs), a new experimental therapy.

The proteins that investigators are targeting in this study are called tumor associated antigens (TAAs). These are cell proteins that are specific to the cancer cell.They either do not show or show up in low quantities on normal human cells. In this study the investigators are targeting five common TAAs called NY-ESO-1, MAGEA4, PRAME, Survivin and SSX. On a different protocol, patients have been treated and so far this treatment has shown to be safe.

Investigators now want to try this treatment in patients with multiple myeloma or if the investigators can arrest the progression of the patient's condition condition (described above) to multiple myeloma.

These TAA-specific CTLs are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the largest safe dose of TAA-specific CTLs, to learn what the side effects are, and to see whether this therapy might help patients with multiple myeloma monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SM)

.

DETAILED DESCRIPTION:
Up to 390 mL (78 teaspoons) of blood will be collected from the patient on one to three occasions over a two month period. Under certain conditions related to the patient's health, the blood may need to be collected using a process called apheresis. Apheresis is the process where blood is passed through a machine that separates out the components of the blood that is needed. The remainder of the blood is then returned to the patient's body.

Investigators will use this blood to grow T cells. They will first grow a special type of cells called dendritic cells which will cause activity in the T cells. Once these are made the investigator will load them with small pieces of protein called peptides taken from the TAAs that they want to target. This helps to train the T cells to kill cells with TAAs on their surface. Then the investigators expand these TAA-specific CTLs.

The cells will be infused by intravenous (IV) infusion into the patient over 10 minutes. The patient may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Initially, two doses of TAA-specific CTLs will be given two weeks apart. The patient's disease will be assessed pre-infusion and then 6 weeks after the second infusion. If after the second infusion there is a decrease in the patient's disease or it remains stable, the patient can receive up to six (6) additional doses of the TAA-specific CTLs at monthly intervals. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

In between the first and second infusions and for 6 weeks after the last infusion, the patient is asked not to receive any other anti-cancer treatments, such as radiation therapy or chemotherapy, with the exception of lenalidomide, thalidomide, pomalidomide, or immune checkpoint inhibitors, such as CTLA4 and/or PD-1/PD-L1 inhibitors. If they do receive any other therapies in-between the first and second infusion of cells, the patient will be taken off treatment and will not be able to receive the second infusion of cells. If the patient bad side effects from the first infusion, he or she will also not be able to receive the second infusion.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose (1 of 3 different levels) of TAA-specific CTLs. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 3 dose levels are studied. If the side-effects are too severe, the dose will be lowered or the TAA-specific CTL infusions will be stopped.

For patients with monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SM), they will receive a fixed dose of TAA-specific CTLs. This dose Was determined based on data obtained from patients who have multiple myeloma and have received these cells.

Medical Tests Before Treatment

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurement of the patient's multiple myeloma, MGUS or SM markers by blood tests and bone marrow biopsy (within 4 weeks before the CTL infusion)
* Measurements of the patient's tumor by routine imaging studies. The investigators will use the imaging study that was used before to follow the patient's tumor: Computerized Tomography (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET/CT), skeletal bone survey. These studies will be done on a case-by-case basis at the descretion of the patient's treating physician.
* Pregnancy test (using a blood sample) if the patient is a female who can have children.

Medical Tests After Treatment:

Patients will receive standard medical tests after their infusion:

* Blood tests to measure blood cells, kidney and liver function.
* Measurement of the patient's multiple myeloma, MGUS or SM markers by blood tests and bone marrow biopsy (at 4-6 weeks and 8-12 weeks post 1st CTL infusion).
* Measurements of your tumor by routine imaging studies. We will use the imaging study that was used before to follow your tumor: Computerized Tomography (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET/CT), skeletal bone survey. These studies will be done on a case-by-case basis at the discretion of your treating physician.

The investigators may request a sample of the patient's previous biopsy (e.g. bone marrow or other tissue) that he or she has had or from a biopsy performed at any time while they are on this study. The sample may be used to measure the multiple myeloma, MGUS or SM in the bone marrow, or for research purposes related to this study.

To learn more about the way the TAA-specific CTLs are working in the patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each infusion, and at Weeks 1, 2, 4 and 6. Afterwards, blood will be collected at 3, 6, 9 and 12 months after the last infusion. The investigators will use this blood to see how long the TAA-specific CTLs last, and to look at the immune response to the cancer. Patients will then be contacted once a year for up to 4 additional years (total of 5 years follow-up) to evaluate their disease response long-term.

ELIGIBILITY:
Procurement Inclusion Criteria

* Any patient, at least 18 yrs old regardless of sex, with a diagnosis of high risk MGUS/smoldering myeloma or patients with a diagnosis of Multiple myeloma after receiving at least one treatment regimen OR
* Any patient, ≥ 18 yrs old regardless of sex with a diagnosis of high risk MGUS (defined as have 2 of the following: 1. Non IgG MGUS, 2. M protein ≥ 1.5 g/dl, 3. Abnormal free light chain ratio (<0.26 for lambda restricted disease or >1.65 for kappa restricted disease) or a diagnosis of smoldering myeloma.
* Patients with life expectancy greater than or equal to 6 weeks.
* Hgb greater than or equal to 7.0 (transfusions allowed).
* Patient able to give informed consent.

Treatment Inclusion Criteria

- Any patient, at least 18 yrs old regardless of sex, with a diagnosis of Myeloma after receiving at least one treatment regimen. If patient has received an autologous or syngeneic SCT they must be >90 days post-transplant (Group A)

OR

Following autologous or syngeneic SCT (as adjuvant therapy) and <90 days post transplant (Group B)

OR

Any patient ≥ 18 yrs old regardless of sex with a diagnosis of high risk MGUS/Smoldering myeloma (definition of high risk MGUS/smoldering myeloma provided in protocol) (Group C)

* Patients with life expectancy greater than or equal to 6 weeks.
* Pulse oximetry of >93% on room air in patients who previously received radiation therapy.
* Patients with a Karnofsky score of greater than or equal to 50.
* Patients with bilirubin less than or equal to 2 times upper limit of normal, AST less than or equal to 3 times upper limit of normal, and Hgb greater than or equal to 7.0 (transfusion allowed).
* Engrafted post transplant (ANC >500) and ANC >500 at the time of infusion if applicable.
* Patients with a creatinine less than or equal to 2x upper limit of normal for age.
* Patients should have been off other investigational therapy for one month prior to entry in this study.
* Patients should have been off conventional therapy for at least 48 hours prior to entry in this study (except for lenalidomide, thalidomide, pomalidomide or immune checkpoint inhibitors such as CTLA4 and/or PD-1/PD-L1 inhibitors)
* Patient able to give informed consent.
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom. Females of child-bearing potential must be willing to utilize one of the more effective birth control methods during the study unless female has had a hysterectomy or tubal ligation.

Procurement Exclusion Criteria

* Patients with severe active infection.
* Patients with active HIV infection at time of procurement (can be pending at the time of blood draw).

Treatment Exclusion Criteria

* Patients with severe active infection.
* Patients receiving systemic corticosteroid within 48 hours of CTL infusion.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-12 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Adverse events | 8 weeks
  To determine the safety of 2 intravenous injections of autologous TAA-specific cytotoxic T-lymphocytes (CTL) in patients with Myeloma as well as those with high risk MGUS/Smoldering myeloma.

SECONDARY OUTCOMES:
Expansion of the CTLs | 1 year
  Information on the expansion of the adoptively transferred tumor-specific CTL will be analyzed for the immunological parameters based on multimer analysis, intracellular cytokine staining and ELIspot assays to assess the frequency of cells secreting γ-IFN using the descriptive statistics such as mean, median, standard deviation at each time point.
Persistence of the CTLs | 1 year
  Information on the persistence of the adoptively transferred tumor-specific CTL will be analyzed for the immunological parameters based on multimer analysis, intracellular cytokine staining and ELIspot assays to assess the frequency of cells secreting γ-IFN using the descriptive statistics such as mean, median, standard deviation at each time point.
Reduction of the Multiple Myeloma | 8 weeks
  Comparison of diagnostic imaging studies from pre-infusion to 6 weeks following the second infusion will be summarized. Frequencies and proportions of responders will be summarized overall and by dose levels if there are enough patients per dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Lulla, MD, Principal Investigator — Baylor College of Medicine/Houston Methodist Hospital
Locations (3):
- United States (3):
  - Harris Health Ben Taub Hospital, Houston, Texas
  - Harris Health Smith Clinic, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No